CLINICAL TRIAL: NCT05727566
Title: Sexual Dysfunction in Patients With Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Yılmaz, MD, asistant prof (MD), Konya Beyhekim Training and Research Hospital
Other Study IDs: KonyaBeyhekimTRH2022
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Sexual Dysfunction; Myofascial Pain Syndrome
Keywords: sexual dysfunction; myofascial pain sydrome; pain
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primer myofascial pain sydrome: pain for at least three months (myofascial pain) reproductive-aged married womens (18-50 years)
  Interventions: Other: visual pain scale (VASpain/fatigue), Beck depression index (BDI), the sexuality-importance score, sexual intercourse frequency
- Healthy controls: Healthy control of reproductive-aged married women with compatible sociodemographic characteristics
  Interventions: Other: visual pain scale (VASpain/fatigue), Beck depression index (BDI), the sexuality-importance score, sexual intercourse frequency

INTERVENTIONS:
Other: visual pain scale (VASpain/fatigue), Beck depression index (BDI), the sexuality-importance score, sexual intercourse frequency — visual pain scale (VASpain/fatigue), Beck depression index (BDI), the sexuality-importance score, sexual intercourse frequency

SUMMARY:
This study evaluates the frequency of sexual dysfunction in women with myofascial pain syndrome and its relationship with clinical parameters.

DETAILED DESCRIPTION:
The frequency of sexual dysfunction in reproductive-aged married women with primary myofascial pain syndrome will be evaluated in a prospective, cross-sectional survey-type study. The medical history of each participant was obtained and they underwent a detailed physical examination. Sociodemographic and clinic characteristics of all participants (age, education, marital status, employment status, family structure, income status, Body Mass Index(BMI), disease duration, number of pregnancies, sleep quality, etc.) were recorded. Pain and fatigue levels of the patients were measured by the visual pain scale (VAS), mood states by the Beck depression index (BDI), sexual function of the participants was assessed by the 0-10 Visual Analog Scale (VAS) to assess the degree of importance of sexuality (the sexuality-importance score). In addition, weekly/monthly sexual intercourse frequency was asked to all participants (patient and control groups). The questionnaires were administered to all participants in a room where they were alone with a female physician, and a suitable environment was provided for the patients to fill out the questionnaire. Patients were assured of the confidentiality of their information. Only questions that were not understood by the patient were explained without guidance.

ELIGIBILITY:
Inclusion Criteria:

* Myofascial pain syndrome (>3 months) was diagnosed in a female.
* Being between the ages of 18 and 50, married, sexually active, and not menopausal
* Volunteering to participate in the study, and being able to communicate easily.

Exclusion Criteria:

* a history of systemic disease (cardiovascular, pulmonary, hepatic, renal, hematological, etc.)
* major psychiatric illness, mental retardation
* uncontrollable respiratory system problems
* endocrine diseases, neurological diseases
* previous hysterectomy or vaginal surgery, a history of sexually transmitted diseases
* urinary or anal incontinence
* limited motion in the upper or lower extremities
* Fibromyalgia
* inflammatory rheumatic diseases (such as rheumatoid arthritis, ankylosing spondylitis, etc.)
* cervical/lumbar radiculopathy or myelopathy
* communication problems
* pregnancy, lactation
* taking estrogen therapy
* use antidepressant, anxiolytic, and antiepileptic drugs
* chronic alcohol users

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 40 patients with primer myofascial pain syndrome and 40 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Sexuality-importance score | 11.05.2022-15.03.2023 (cross-sectional)
  Sexual function of the participants was assessed by the 0 (never mind)-10(very important) Visual Analog Scale (VAS) to assess the degree of importance of sexuality.
The frequency of sexual intercourse | 11.05.2022-15.03.2023 (cross-sectional
  Weekly/monthly sexual intercourse frequency was asked of all participants.

SECONDARY OUTCOMES:
Visual analog scale (VAS pain/fatigue) | 11.05.2022 - 15.03.2023 (cross-sectional)
  All participants were assessed in terms of pain and fatigue levels by means of a visual analogue scale of 0-10 cm (VAS).
Beck depression index (BDI) | 11.05.2022 - 15.03.2023 (cross-sectional)
  In the assessment of depression severity, the Turkish version of the 21-item Beck Depression Inventory (BDI) was used, which is one of the most common psychometric tests used and a value of 0 to 3 is assigned for each answer to each item.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Yılmaz, asist. prof, Study Chair — Konya Beyhekim Training and Research Hospital, Konya, Turkey
Locations (1):
- University of Health Sciences, Konya Beyhekim Training and Research Hospital, Department of Physical Medicine and Rehabilitation, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yilmaz H, Yilmaz SD, Polat HA, Salli A, Erkin G, Ugurlu H. The effects of fibromyalgia syndrome on female sexuality: a controlled study. J Sex Med. 2012 Mar;9(3):779-85. doi: 10.1111/j.1743-6109.2011.02619.x. Epub 2012 Jan 12. PMID 22240036
- [Derived] Yilmaz R, Karpuz S, Akdere E, Yilmaz H. Evaluation of sexual dysfunction in females with neck and upper back myofascial pain syndrome: a cross-sectional study. Rheumatol Int. 2023 Sep;43(9):1723-1732. doi: 10.1007/s00296-023-05359-6. Epub 2023 Jun 9. PMID 37294458